CLINICAL TRIAL: NCT02942147
Title: Comparison of the Efficacy of Conventional Radiofrequency, Pulse Radiofrequency, and TENS Therapies for Lumbar Facet Joint Pain: A Single-blind Randomized Controlled Trial
Brief Title: Conventional Radiofrequency, Pulse Radiofrequency, and TENS for Lumbar Facet Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Sibel Eyigor, Prof, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIP
Record Dates: First submitted 2016-10-14; First posted 2016-10-21 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Transcutaneous Electric Nerve Stimulation; Congresses as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- conventional radiofrequency therapy (Active Comparator): In the conventional radiofrequency method applied to Group 1 patients, the targeted facet joints were marked while the fluoroscope was in antero-posterior position.
  Interventions: Procedure: Conventional or Pulse Radiofrequency
- conventional TENS (Active Comparator): Group 2 patients were administered TENS therapy 30 minutes a day for 15 days at the outpatient physiotherapy unit of the Physiotherapy and Rehabilitation Department. The TENS therapy was applied in the form of conventional TENS subtype with 80-100 Hz frequency by placing four electrodes on the region where the pain was most intense.
  Interventions: Device: TENS
- pulse radiofrequency therapy (Active Comparator): In the pulse radiofrequency method applied to Group 3 patients, the targeted facet joints were marked while the fluoroscope was in antero-posterior position.
  Interventions: Procedure: Conventional or Pulse Radiofrequency

INTERVENTIONS:
Device: TENS — Group 2 patients were administered TENS therapy 30 minutes a day for 15 days at the outpatient physiotherapy unit of the Physiotherapy and Rehabilitation Department. The TENS therapy was applied in the form of conventional TENS subtype with 80-100 Hz frequency by placing four electrodes on the region where the pain was most intense.
  Arms: conventional TENS
Procedure: Conventional or Pulse Radiofrequency — In the radiofrequency method applied to Group 1 and Group 3 patients, the targeted facet joints were marked while the fluoroscope was in antero-posterior position. During this marking, the fluoroscope was directed towards cephal or caudal so that at whatever level the median ramus block was to be involved the endplate of that vertebra would become a straight line. The connection point of the superior articular protrusion was marked on the fluoroscope using the transverse process and the intervention was applied with a 22G, 10-cm radiofrequency cannula with 0.5 cm active tip in a way that bone contact was established through the tunneled vision technique. The intervention was completed after the radiofrequency procedure was applied at four levels.
  Arms: conventional radiofrequency therapy; pulse radiofrequency therapy

SUMMARY:
Objective: The objective of this study is to compare the efficacy of TENS (transcutaneous electrical nerve stimulation) therapy with those of the conventional radiofrequency and pulse radiofrequency therapies.

Design: A single-blind randomized controlled trial

Setting: An outpatient physical therapy and rehabilitation clinic

Subjects: The study included 60 patients who presented with a complaint of chronic low back pain prevailing at least for 3 months and who were diagnosed with facet joint syndrome.

Interventions: The patients were randomized into 3 groups so that Group 1 (n: 20) patients would receive conventional radiofrequency therapy, Group 2 (n: 20) patients conventional TENS procedure for 15 days and Group 3 (n: 20) patients pulse radiofrequency therapy.

Main measures: The patients were assessed before treatment, and at month 1 and 6 for pain (visual analogue scale), disability (Oswestry Disability Index), lumbar movements (hand-floor distance), functional status (20-meter walking times, 6-min walking distances), quality of life (Short Form 36), and depression (Beck Depression Inventory).

DETAILED DESCRIPTION:
Patient selection

The study included patients who presented to the outpatient clinics of these units with the complaint of chronic low back pain prevailing for at least 3 months that had not responded to previous medical treatment. Medical history were obtained from the patients and their low back and lower extremity musculoskeletal systems and neurologic systems were examined. Patients were assessed using their two-way lumbar X-rays taken within the last 1 year and lumbar magnetic resonance imaging outcomes. After all these examinations and assessments, the patients who were excluded from the study consisted of those who had a coagulation disorder, a history of malignity, a mental disorder, a psychiatric disorder, pregnancy, prior low back surgery, a history of TENS or radiofrequency procedure at their low back region within the last 1 year, an advanced (grade 3-4) spondylolisthesis defect in their lumbar vertebrae, an extruded and sequestrated disk hernia or a spinal narrow canal in their magnetic resonance imaging, a cauda equine syndrome or advanced paresis, an examination finding suggesting radiculopathy with pain noticeably extending under the knee, a history of systemic inflammatory disease, an advanced cardiac deficiency and a diagnosis of pulmonary disease. In the light of the medical history, examination findings and other tests, the patients who were thought to have facet joint syndrome and who did not meet any of the exclusion criteria above were informed about the study and treatment procedures.

The patients who agreed to receive the treatment based on the information given to them were administered a diagnostic test dose at the operating room of the Algology Division to confirm whether the present pain was associated with the facet syndrome meeting the inclusion criteria. This diagnostic procedure involved injection of 0.4 cc of bupivacaine under fluoroscopy to the median of dorsal ramus that enable innervation of lumbar facet joints. The patients whose pain receded more than 50% after this administration of a test dose and who met the other two inclusion criteria, visual analogue scale pain level >3 and 18-75 years of age, were included in the study.

The patients included in the study were informed both in writing and verbally about the purpose and length of the study, the way of implementing it, and possible side effects and problems that can arise. Patients signed the "subject informed consent form" and local ethics committee approval was obtained.

Intervention

The study was designed as a prospective, randomized, single-blind study. While the patients had knowledge of what the treatment was, the physician who made the assessments before and after the treatment did not know what treatment the patient received. The randomization template obtained from www. randomizer.org was used to randomize the patients.

The patients were divided into three groups according to the randomization template. Group 1 patients (n: 20) were administered the conventional radiofrequency procedure, Group 2 patients (n: 20) the TENS (transcutaneous electrical nerve stimulation) procedure and Group 3 patients (n: 20) the pulse radiofrequency procedure.

For the purposes of safety and drug administration, vascular access was established in the operating room of the Algology Division in both the patients who would undergo a diagnostic test and those who would receive the actual treatments, the conventional and pulse radiofrequency therapies. The patients were laid in supine position; their procedural sites were sterilized and covered with a sterile cover. All procedures were carried out under fluoroscopy.

In the conventional radiofrequency method applied to Group 1 patients, the targeted facet joints were marked while the fluoroscope was in antero-posterior position. During this marking, the fluoroscope was directed towards cephal or caudal so that at whatever level the median ramus block was to be involved the endplate of that vertebra would become a straight line. Afterwards, the fluoroscope was brought to oblique 45 degrees on facets L4-5 and L5-S1 and 30 degrees on the upper facets. The connection point of the superior articular protrusion was marked on the fluoroscope using the transverse process and the intervention was applied with a 22G, 10-cm radiofrequency cannula with 0.5 cm active tip in a way that bone contact was established through the tunneled vision technique. The intervention was completed after the conventional radiofrequency procedure was applied at four levels (L2-L3, L3-L4, L4-L5 and L5-S1) at 80 degrees for 1 minute at each level.

Group 2 patients were administered TENS therapy 30 minutes a day for 15 days at the outpatient physiotherapy unit of the Physiotherapy and Rehabilitation Department. The TENS therapy was applied in the form of conventional TENS subtype with 80-100 Hz frequency by placing four electrodes on the region where the pain was most intense.

In the pulse radiofrequency method applied to Group 3 patients, the targeted facet joints were marked while the fluoroscope was in antero-posterior position. During this marking, the fluoroscope was directed towards cephal or caudal so that at whatever level the median ramus block was to be involved the endplate of that vertebra would become a straight line. Afterwards, the fluoroscope was given an oblique position 45 degrees at L4-5 and L5-S1levels and 30 degrees at the upper levels. The connection point of the vertebral corpus was marked on the fluoroscope using the transverse process and the intervention was applied with a 22G, 10-cm radiofrequency cannula with 0.5 cm active tip in a way that bone contact was established through the tunneled vision technique. The intervention was completed after a 45-V pulse radiofrequency procedure was applied at 4 levels (L2-L3, L3-L4, L4-L5 and L5-S1) at 42oC for 4 minutes at each level.

Additionally, all 3 groups of patients were given a home exercise program in the form of lumbar range of motion and lumbar isometric exercises except extensional and rotational movements to be performed at least twice a week throughout the follow-up period. The patients were phoned every week to encourage them to comply with the exercise program.

ELIGIBILITY:
Inclusion Criteria:

* The study included patients who presented to the outpatient clinics of these units with the complaint of chronic low back pain prevailing for at least 3 months that had not responded to previous medical treatment

Exclusion Criteria:

The patients who were excluded from the study consisted of those who had:

* coagulation disorder
* history of malignity
* mental disorder
* psychiatric disorder
* pregnancy
* prior low back surgery
* advanced (grade 3-4) spondylolisthesis defect
* extruded and sequestrated disk hernia
* spinal narrow canal
* cauda equine syndrome
* history of systemic inflammatory disease
* advanced cardiac deficiency
* diagnosis of pulmonary disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Change-Visual Analogue Scale | Pre-treatment, 1 month, 6 month

SECONDARY OUTCOMES:
Change-Oswestry Disability Index | 0 month, 1 month, 6 month
Change-Short Form 36 | 0 month, 1 month, 6 month
Change-Beck Depression Inventory | 0 month, 1 month, 6 month

IPD SHARING:
Plan to Share IPD: Undecided